CLINICAL TRIAL: NCT06941896
Title: Study of the Effect of the Atalante Exoskeleton (Wandercraft) on Autonomy in Individuals With Paraplegia Undergoing Rehabilitation (Standing and Walking): A Prospective Uncontrolled Study in a Controlled Environment to Demonstrate Its Physical and Psychosocial Utility.
Brief Title: Effect of the Atalante Exoskeleton on Standing and Walking in Individuals With Paraplegia: A Prospective Controlled-Environment Study in a Rehabilitation Context
Acronym: APPEX
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Principal Investigator, Eric Pantera, Principal Investigator, Medical Doctor, Specialist in Physical and Rehabilitation Medicine, CHU de Nîmes; Research Affiliate, Euromov Laboratory, University of Montpellier, Centre Hospitalier Universitaire de Nīmes
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2016-A01221-50
Record Dates: First submitted 2025-04-01; First posted 2025-04-24 (Actual); Last update posted 2025-04-24 (Actual); Status verified 2025-04

CONDITIONS: Paraplegia, Complete
Keywords: exoskeleton; Atalante; paraplegia; rehabilitation; safety
MeSH Terms: conditions — Paraplegia

STUDY DESIGN:
Intervention Model Description: All participants will receive the same intervention: the use of the Atalante exoskeleton for assisted standing and walking during rehabilitation. There is no control group.
Masking Description: No blinding was applied, as all participants and investigators were aware of the intervention during the sessions.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Exosquelette Atalante (Experimental)
  Interventions: Device: Use of the Atalante Exoskeleton

INTERVENTIONS:
Device: Use of the Atalante Exoskeleton — Assisted verticalization (sit-to-stand transition)
  Orthostatic stabilization (unsupported standing posture)
  Assisted locomotion (stabilized walking)

SUMMARY:
This clinical study aims to evaluate the feasibility, safety, and acceptability of the Atalante robotic exoskeleton, developed by Wandercraft, within a functional rehabilitation protocol for individuals with complete paraplegia. Unlike re-education, which focuses on restoring impaired functions, rehabilitation seeks to promote long-term autonomy despite persistent impairments.

The study would involve adult participants with complete spinal cord injury-induced paraplegia. Each participant would follow an intensive program of 60 sessions over six weeks, including phases of verticalization, postural stabilization, and assisted locomotion. The protocol would include three evaluation domains: (1) biomedical safety (orthostatic tolerance, adverse events, metabolic load), (2) techno-functional usability (setup time, technical incidents), and (3) user-perceived trust (comfort, sense of safety, satisfaction).

The primary objective would be to determine whether the Atalante exoskeleton can be safely and repeatedly used by individuals with complete paraplegia without requiring manual support. The study would also aim to identify potential barriers to its integration into an intensive rehabilitation protocol. The expected outcomes could guide clinical practices and help define optimal inclusion criteria for the safe and effective use of this technology.

DETAILED DESCRIPTION:
Background and Rationale Complete paraplegia, resulting from spinal cord injury, is a major neurological condition involving irreversible loss of lower limb function. Given the limitations of neuromotor re-education in such contexts, rehabilitation aims to restore autonomy and social participation by leveraging residual capacities and assistive technologies. Robotic exoskeletons represent a promising technological innovation in this domain by offering assisted locomotion that compensates for loss of mobility.

Among these devices, Atalante (Wandercraft, Paris, France) is a next-generation, self-stabilizing exoskeleton designed to enable dynamic walking without manual support, through a fully motorized lower limb system. Unlike conventional devices that require crutches or canes, Atalante provides active stabilization, offering new perspectives in terms of autonomy, safety, comfort, and quality of life.

While the potential benefits of exoskeletons in motor recovery have been explored, their use in a functional rehabilitation context remains under-investigated. This project therefore aims to evaluate the Atalante exoskeleton as an assistive tool for autonomy within a structured intensive protocol in a safe clinical environment.

Primary Objective To evaluate the feasibility, safety, and acceptability of intensive use of the Atalante exoskeleton in a functional rehabilitation context among adults with chronic complete paraplegia.

Secondary Objectives To determine the number of sessions required to reach operational familiarization with the exoskeleton.

To describe technical incidents and their impact on comfort and perceived safety.

To assess the energy cost of assisted locomotion.

To identify potential bone contraindication criteria based on bone mineral density (T-score).

To measure the evolution of user satisfaction throughout the protocol.

Investigational Device: Atalante Exoskeleton

The Atalante exoskeleton is an active robotic system with 12 powered degrees of freedom symmetrically distributed across both lower limbs (3 at the hip, 1 at the knee, 2 at the ankle). It enables:

Biomimetic joint movements,

Active postural control,

Self-stabilized dynamic walking without external support.

Its hybrid control system (continuous/discrete time) is based on Hybrid Zero Dynamics algorithms, which optimize movement trajectories and ensure real-time dynamic balance. The user interface allows switching between multiple modes (sit-to-stand, walk, stop) via remote control. Inertial sensors, angular encoders, and pressure sensors detect the user's intention to move.

Study Design Type: Prospective, single-center, longitudinal, non-randomized study.

Intervention duration: 6 weeks (60 sessions per participant).

Location: Centre de Médecine Physique et Réadaptation APAJH, Pionsat (France).

Safety setup: Overhead rail system with active fall protection, non-interfering with device operation.

Population Participants will be adults with complete paraplegia (ASIA A), lesion level ≤ T6, with stabilized spinal cord injury. They must present anthropometric parameters compatible with the exoskeleton (height, weight, joint mobility). Selection will be based on strict eligibility criteria (see "Eligibility" section).

Intervention Protocol

Each participant will undergo:

2 sessions/day, 5 days/week for 6 weeks.

Each session includes:

Assisted verticalization (sit-to-stand),

Orthostatic stabilization (upright stance without support),

Assisted locomotion (stabilized walking).

Sessions will be supervised by trained professionals. A session will be considered valid if the participant completes a 40-meter round trip without incident. The intensity of the program is designed to simulate realistic sustained home use.

Evaluation Domains

1. Biomedical Safety

   Monitoring of adverse events (major and minor): fractures, skin abrasions, orthostatic hypotension, pain.

   Metabolic analysis (VO₂, cost of transport, perceived exertion via Borg scale) during sessions 21 and 60.

   Exploratory contraindication: T-score < -3.5 at the hip (severe osteoporosis).
2. Techno-Functional Usability

   Donning and doffing times (sessions 1 to 60),

   Number and type of technical incidents: unexpected stops, deviations, backward perturbations, software bugs.

   Functional familiarization assessment (Elbow Curve method).
3. Perceived Confidence and Acceptability

Session-end assessments via:

Visual analog scales (VAS): general comfort, thoracic harness comfort, safety while standing, walking, and during transitions.

QUEST 2.0 questionnaire at the end of the protocol.

Data Analysis Methodology Quantitative data will be expressed as means ± standard deviation or medians (interquartile ranges).

Intra-subject pre/post comparisons: Student's t-test for parametric data, Wilcoxon test otherwise.

Longitudinal follow-up: progression curves for donning time, technical incidents, and VAS scores.

Effect size and significance thresholds: p < 0.05; 95% confidence intervals.

Ethics The study will be conducted in accordance with the principles of the Declaration of Helsinki. It has received approval from the Ethics Committee (CPP) and the French Medicines Agency (ANSM). All participants will sign informed consent. French CPP : 2016-A01221-50.

Expected Outcomes

The results of this study could:

Confirm the relevance of Atalante in a functional rehabilitation approach,

Provide practical recommendations for safe clinical use,

Prepare future multicenter studies in real-life environments (home, urban spaces),

Contribute to the development of eligibility criteria for prescribing exoskeletons as assistive mobility devices.

ELIGIBILITY:
Inclusion Criteria:

* Complete spinal cord injury (ASIA A classification)
* Lesion level at or below T6
* Injury occurred more than 6 months prior to enrollment (chronic/stabilized injury)
* Ability to maintain upright posture without symptomatic orthostatic hypotension
* Joint range of motion compatible with wearing the exoskeleton
* Anthropometric dimensions compatible with the device, including:
* Body weight less than 90 kg

Exclusion Criteria:

* Spasticity greater than 3 on the Modified Ashworth Scale
* Joint limitations incompatible with exoskeleton use
* Spinal instability
* Cognitive or psychiatric disorders affecting protocol adherence
* Recent dermatological conditions
* History of fragility fractures in the lower limbs within the past 2 years
* Presence of 5 or more fracture risk factors according to Craven et al., including:

  * Injury older than 10 years
  * Thoracic-level lesion
  * Absence of regular weight-bearing activity
  * Low spasticity
  * Body Mass Index (BMI) < 20
* Cardiopulmonary contraindications to physical effort
* Pregnancy or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2019-09 (Actual); Study Completion 2019-09 (Actual)

PRIMARY OUTCOMES:
Adverse events related to the use of the Atalante exoskeleton | At each session, through study completion (6 weeks total)
  Evaluation of biomedical safety through systematic recording of adverse events (serious and non-serious) occurring during the training program, including but not limited to: fractures, dermabrasions, orthostatic hypotension, joint or muscle pain.

SECONDARY OUTCOMES:
Evolution of oxygen consumption during assisted locomotion | Session 21 (week 3) and session 60 (week 6)
  Measurement of oxygen consumption (VO₂) during a 6-minute walk test using the Atalante exoskeleton. Results are expressed in mL O₂/kg/m.
Evolution of transport cost during assisted locomotion | Session 21 (week 3) and session 60 (week 6)
  Measurement of transport cost calculated from oxygen consumption data during a 6-minute walk test with the Atalante exoskeleton.
  Unitless or specify your formula (e.g., mL O₂/kg/m)
Evolution of perceived exertion during assisted locomotion | Session 21 (week 3) and session 60 (week 6)
  Assessment of perceived exertion using the Borg Rating of Perceived Exertion (RPE) scale after a 6-minute walk test with the Atalante exoskeleton. The Borg scale ranges from 0 (no exertion) to 10 (maximal exertion). Higher scores indicate greater perceived exertion. Units:
  Points on the Borg RPE scale (0-10)
Perceived general comfort during use of the Atalante exoskeleton | At each session, through study completion (6 weeks total)
  Evaluation of general comfort using a Visual Analog Scale (VAS) during sit-to-stand, standing, and walking with the Atalante exoskeleton. The VAS ranges from 0 mm (no discomfort) to 100 mm (maximal discomfort). Lower scores indicate better comfort.
  Units: mm on VAS (0-100 mm)
Perceived thoracic comfort during use of the Atalante exoskeleton | At each session, through study completion (6 weeks total)
  Evaluation of thoracic comfort using a Visual Analog Scale (VAS) during sit-to-stand, standing, and walking with the Atalante exoskeleton. The VAS ranges from 0 mm (no discomfort) to 100 mm (maximal discomfort). Lower scores indicate better thoracic comfort.
  Units: mm on VAS (0-100 mm)
Perceived feeling of safety during use of the Atalante exoskeleton | At each session, through study completion (6 weeks total)
  Evaluation of participants' perceived safety using a Visual Analog Scale (VAS) during sit-to-stand, standing, and walking with the Atalante exoskeleton. The VAS ranges from 0 mm (no feeling of safety) to 100 mm (maximal feeling of safety). Higher scores indicate greater perceived safety.
  Units: mm on VAS (0-100 mm)
Participant satisfaction with the Atalante exoskeleton assessed by the Quebec User Evaluation of Satisfaction with Assistive Technology (QUEST 2.0) scale | At study completion (week 6)
  Evaluation of overall satisfaction with the Atalante exoskeleton using the Quebec User Evaluation of Satisfaction with Assistive Technology (QUEST 2.0) scale. This standardized questionnaire includes 8 items rated from 1 (not satisfied at all) to 5 (very satisfied), assessing comfort, safety, ease of use, durability, effectiveness, aesthetics, and adjustability. Higher scores indicate greater satisfaction. Units:
  Points on QUEST 2.0 scale (1-5 per item; total score range: 8-40)
Change in donning and doffing time for the exoskeleton | At each session, through study completion (6 weeks total)
  Measurement (in seconds) of time required to put on and remove the exoskeleton at each session. Analysis of progression in technical handling over time.
Frequency and types of technical incidents | At each session, through study completion (6 weeks total)
  Systematic recording of technical incidents (minor and major), including unexpected shutdowns, software errors, trajectory deviations, and other anomalies. Data correlated with participant perception of safety and session interruptions.
Number of sessions required for functional familiarization with the exoskeleton | Through study completion (up to 6 weeks)
  Estimation of the number of training sessions needed for each participant to reach a performance plateau in donning and doffing the Atalante exoskeleton. The plateau is defined via curve inflection analysis using the Elbow Method. Units: Number of sessions

CONTACTS AND LOCATIONS:
Locations (1):
- CMPR APAJH Pionsat, Pionsat, Auvergne, France

IPD SHARING:
Plan to Share IPD: No
The sharing of individual participant data is not planned at this stage due to the exploratory nature of the study and the limited sample size. However, anonymized data could be made available upon a justified request, subject to approval by the ethics committee and the sponsor, within the framework of a scientific collaboration or future meta-analyses